CLINICAL TRIAL: NCT03720236
Title: Behavior of Peri-implant Tissues in BLX® Implants Placed on Mature Scarred Bone
Brief Title: Peri-implant Tissues in BLX® Implants
Acronym: BLX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Manohay Dental SAU (Unknown)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-2018-05
Record Dates: First submitted 2018-10-05; First posted 2018-10-25 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Dental Implant Failed; Dental Prosthesis Failure
Keywords: dental implant; immediate loading; periimplant tissues
MeSH Terms: interventions — O,O-diisopropyl-S-benzylthiophosphate; Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Full preparation (Experimental): Group A: the complete milling protocol indicated by the manufacturer for the 3.75x10 mm BLX implant will be performed.
  Interventions: Procedure: Implant bed preparation protocol
- Partial preparation (Experimental): Group B: the partial / under milling protocol for the 3.75x10 mm implant, indicated by the manufacturer, will be carried out.
  Interventions: Procedure: Implant bed preparation protocol
- Deferred loading (Experimental): Code 2: for implants with this random code, the prosthetic prosthesis SRA of 2.5 mm and its corresponding healing plug of 5.1 mm will be placed. Impressions will be taken at 6 weeks to place the provisional prosthesis at 8 weeks. At 6 months the final impressions will be taken for the definitive load.
  Interventions: Procedure: Implant loading
- Immediate load (Experimental): The code 1: to the implants with this random code, the prosthetic prosthesis SRA of 2.5 mm and its corresponding healing plug of 5.1 mm will be placed. The impression will be made in the same surgery and the placement of the provisional prosthesis before 7 days. At 6 months the final impressions will be taken for the definitive load.
  Interventions: Procedure: Implant loading

INTERVENTIONS:
Procedure: Implant bed preparation protocol — This is the first surgical phase, we prepare the implant bed by using different increasing size drills.
  Other Names: IBP
  Arms: Full preparation; Partial preparation
Procedure: Implant loading — This is the second phase, based on prosthetic procedures, to design the crown over the dental implant
  Other Names: IL
  Arms: Deferred loading; Immediate load

SUMMARY:
This is a randomized triple-blind clinical trial to evaluate the behavior of peri-implant tissues (bone and soft tissues) in BLX implants loaded early or delayed and with different surgical milling protocols. To this end, 40 BLX implants with a diameter of 3.75x10 will be placed in areas of mature bone scarred after extraction. They will be divided into 2 study groups, and these in turn into two subgroups. Group A: complete milling, Group B: partial milling. Each group will be assigned with code 1: early load and code 2: deferred load. Clinical and radiological parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients without systemic pathology
* Adult of age who agree to be part of the study and sign the informed consent.
* Patients smoking less than 5 cigarettes / day,
* Patients not being completely edentulous
* Unitary / multiple absences in the area posterior with or without free ends to distal, maxillary or mandibular that do not require regenerative techniques
* Area of mature bone healed at least 6 months post-extraction.
* The minimum torque for early loading will be 25 N. The placement of the implant will be mechanical up to 40 N maximum and manually finished with a surgical dynamometer.
* The placement of the abutment will be at a minimum of 25 N, in case the primary stability of the implant allows it, it will be placed at 35 N.
* The placement of the implant must always be 4 mm below the future gingival margi

Exclusion Criteria:

* Immunosuppressed patients
* Aesthetic edentulous areas of 13-23 and 33-43
* Smokers of more than 5 cigarettes
* Implants with a lower torque whose will be submerged with a screw and a protocol will be followed in 2 phases, being discarded from the study.
* Index of bleeding greater than 30%
* Patients with less than 2 mm of keratinized gingiva
* Implants with ISQ index <55
* When a margin of 1 mm safety cannot be assumed to the inferior dental nerve

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Primary stability of implants and peri-implant tissues | 12 months
  Randomly and following the inclusion and exclusion criteria, the implants will be placed with the normal preparation protocol (n = 20) and with the preparation protocol with under-fresh (n = 20). We will evaluate the immediate post-surgical stability of implants and peri-implant tissues through the Ostell system, based on the resonance frequency analysis (RFA). The implant stability quotient (ISQ) is the value on a scale that indicates the level of stability and osseointegration in dental implants. The scale ranges from 1 to 100, with higher values indicating greater stability. The acceptable stability range lies between 55-85 ISQ

SECONDARY OUTCOMES:
Basal Peri-implant tissue level: implant stability | 1 day
  Randomly and following the inclusion and exclusion criteria, the implants will be placed with the normal preparation protocol (n = 20) and with the preparation protocol with under-fresh (n = 20). We will load the crowns in two different groups, code 1: loading the implants before 7 days after surgery; code 2: before 8 weeks after implant surgery. We will evaluate the stability at different moments, 8 weeks, 6 months and 12 months.The implant stability quotient (ISQ) is the value on a scale that indicates the level of stability and osseointegration in dental implants. The scale ranges from 1 to 100, with higher values indicating greater stability. The acceptable stability range lies between 55-85 ISQ. ISQ values are obtained using resonance frequency analysis (RFA).
Basal Radiological Bone Implant level | 1 day
  At the moment of placing the implant a periapical radiography will be performed, considering this measure the basal radiological bone level (distance from the neck of the implant to the most crestal level of the alveolar bone). We will calculate the difference between the basal measure and the future measurements.
Basal Peri-implant tissue level: probing depth | 1 day
  At the moment of placing the implant, clinical variables will be evaluated: depth of probing (distance from the peri-implant margin to the most depth of the peri-implant sulcus). This will be the basal measure of the implant stability and peri-implant tissue levels. We will calculate the difference between the basal measure and the future measurements.
Radiological bone implant stability | 6 weeks
  After the implantation, we´ll load the temporary prostheses in two different moments, 7 days or 8 weeks depending of the aleatory coding. We will evaluate the bone level stability at 6 weeks in both groups. The bone stability will be measured as a difference between de basal bone level and the actual one in mm.
Peri-implant tissue stability: probing depth | 6 weeks
  After the implantation, we´ll load the temporary prostheses in two different moments, 7 days or 8 weeks depending of the aleatory coding. We will evaluate the peri-implant tissue stability by measuring the probing depth or just in case, the recession of the gingival margin. The stability will be gave by the differences between both measures, basal and actual in mm.
Peri-implant tissue stability: ISQ | 6 weeks
  After the implantation, we´ll load the temporary prostheses in two different moments, 7 days or 8 weeks depending of the aleatory coding. We will evaluate the peri-implant tissue stability by measuring the ISQ through RFA. The stability will be gave by the differences between both measures, basal and actual.
Clinical tissue levels of definitive prostheses: probing depth | 6 months
  The final or definitive prostheses will be inserted in all groups at 6 months. At this time, we will measure the clinical probing depth, comparing with previous measurements.
Clinical tissue levels of definitive prostheses: ISQ | 6 months
  The final or definitive prostheses will be inserted in all groups at 6 months. At this time, we will measure the implant stability through RFA, comparing with previous measurements.
Radiological tissue levels of definitive prostheses: bone implant level | 6 months
  The final or definitive prostheses will be inserted in all groups at 6 months. At this time, we will measure the bone implant level by measuring the distance from de implant neck to the most apical inserted bone, comparing simultaneously with previous measurements.

OTHER OUTCOMES:
Long-term evaluation of definitive prostheses | 12 months
  After 6 months of loading of final ceramic restoration, we will evaluate the differences of clinical (mm of probing depth, ISQ implant stability) and radiological aspects (bone implant level in mm calculated from the neck to the actual bone level, comparing on the basal, the intermediate, and final values.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Perez Sayans, PhD, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Mario Pérez Sayáns, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will anonymize and categorize the clinical and radiological data of the patients to share the information with the other researchers of the group (n=9)
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From the beginning to sex month after finishing the study
Access Criteria: Under request

REFERENCES:
- See also: GI-1319 — http://imaisd.usc.es/grupoficha.asp?idpersoatipogrupo=75189&i=es&s=-2-26-148